CLINICAL TRIAL: NCT02459106
Title: Effect of AT-derived miRNA on the Biology and Insulin Sensitivity of Skeletal Muscle in Humans
Acronym: miRNA
Status: Completed | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TRIMDFH 729828
Record Dates: First submitted 2015-05-22; First posted 2015-06-01 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: micro-RNA; insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Muscle and adipose tissue biopsies will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy lean insulin-sensitive individuals: This group will be studied by measuring the adipose tissue miRNA release, adipose tissue-released miRNA will be profiled, and these effects will be examined.
- Obese insulin-resistant individuals: This group will be studied by measuring the effect of adipose tissue-release miRNA on skeletal muscle biology and insulin sensitivity, adipose tissue-released miRNA will be profiled, and these effects will be examined on obese insulin-resistant individuals on skeletal muscle biology and insulin sensitivity.

SUMMARY:
The purpose of this study is examine the effect of fat tissue-released miRNA on skeletal muscle and if abnormal fat tissue-released miRNA contributes to insulin resistance in obese individuals. This information will be important for our understanding of how the body's sugar metabolism is regulated and why people who are obese become insulin resistant and are more likely to develop type 2 diabetes.

DETAILED DESCRIPTION:
Study Objectives:

1. To establish and optimize the methodology for measuring adipose tissue miRNA release.
2. To establish and optimize the methodology for measuring the effect of adipose tissue-released miRNA on skeletal muscle biology and insulin sensitivity.
3. To profile adipose tissue-released miRNA in lean insulin-sensitive and obese insulin-resistant healthy individuals.
4. To examine the effects of adipose tissue-released miRNA from lean insulin-sensitive individuals and obese insulin-resistant individuals on skeletal muscle biology and insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate meaningfully with the investigator and legally competent to provide informed written consent
* 18-65 years of age
* BMI of 20-25 kg/m2 (lean subjects); 30-35 kg/m2 (obese subjects)
* Stable body weight (< 3 kg change in the last 8 weeks)
* homeostatic model assessment (HOMA)-insulin resistance <2.7 if lean; homeostatic model assessment (HOMA)-insulin resistance ≥2.7 if obese

Exclusion Criteria:

* Lactation or pregnancy, current and/or within last 6 months, per participant's report
* Female subjects postmenopausal
* Cardiovascular disease (unstable angina, myocardial infarction or coronary revascularization within 6 months)
* Liver disease (AST or ALT(alanine aminotransferase)>2.5 times the upper limit of normal)
* Kidney disease (creatinine >1.6 mg/dl)
* Anemia (hemoglobin <12 g/dl in men, <11 g/dl in women)
* Thyroid dysfunction (abnormal TSH)
* HbA1c ≥6.5%
* Uncontrolled hypertension (systolic BP>160 mmHg, diastolic BP>100 mmHg)
* History of coagulopathies
* History (within the last 5 years) or presence of malignancy, (skin cancers, with the exception of melanoma, may be acceptable)
* Current or history of drug abuse or alcohol abuse (>2 drinks/day)
* Prior treatment (within last 3 months) with systemic glucocorticoids (>2 weeks), beta-blockers, drugs for weight loss, niacin or fibrates
* History of HIV, active Hepatitis B or C, or Tuberculosis (participant reported)
* Smoke > 5 cigarettes per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy obese insulin-resistant individuals Healthy lean insulin-sensitive individuals
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2017-01-24 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Levels of miRNA will be measured as well as the adipose tissue specific miRNA. | 4 weeks
  The effect of miRNA released by adipose tissue from lean insulin-sensitive and from obese insulin-resistant individuals on skeletal muscle biology and insulin signaling.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pratley, MD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

REFERENCES:
- [Background] Coppack SW, Jensen MD, Miles JM. In vivo regulation of lipolysis in humans. J Lipid Res. 1994 Feb;35(2):177-93. PMID 8169522
- [Background] Trayhurn P. Endocrine and signalling role of adipose tissue: new perspectives on fat. Acta Physiol Scand. 2005 Aug;184(4):285-93. doi: 10.1111/j.1365-201X.2005.01468.x. PMID 16026420
- [Background] Flier JS. Obesity wars: molecular progress confronts an expanding epidemic. Cell. 2004 Jan 23;116(2):337-50. doi: 10.1016/s0092-8674(03)01081-x. PMID 14744442
- [Background] Xie H, Sun L, Lodish HF. Targeting microRNAs in obesity. Expert Opin Ther Targets. 2009 Oct;13(10):1227-38. doi: 10.1517/14728220903190707. PMID 19650761
- [Background] Karbiener M, Fischer C, Nowitsch S, Opriessnig P, Papak C, Ailhaud G, Dani C, Amri EZ, Scheideler M. microRNA miR-27b impairs human adipocyte differentiation and targets PPARgamma. Biochem Biophys Res Commun. 2009 Dec 11;390(2):247-51. doi: 10.1016/j.bbrc.2009.09.098. Epub 2009 Oct 2. PMID 19800867
- [Background] Kim SY, Kim AY, Lee HW, Son YH, Lee GY, Lee JW, Lee YS, Kim JB. miR-27a is a negative regulator of adipocyte differentiation via suppressing PPARgamma expression. Biochem Biophys Res Commun. 2010 Feb 12;392(3):323-8. doi: 10.1016/j.bbrc.2010.01.012. Epub 2010 Jan 7. PMID 20060380
- [Background] Ortega FJ, Moreno-Navarrete JM, Pardo G, Sabater M, Hummel M, Ferrer A, Rodriguez-Hermosa JI, Ruiz B, Ricart W, Peral B, Fernandez-Real JM. MiRNA expression profile of human subcutaneous adipose and during adipocyte differentiation. PLoS One. 2010 Feb 2;5(2):e9022. doi: 10.1371/journal.pone.0009022. PMID 20126310
- [Background] Sun L, Xie H, Mori MA, Alexander R, Yuan B, Hattangadi SM, Liu Q, Kahn CR, Lodish HF. Mir193b-365 is essential for brown fat differentiation. Nat Cell Biol. 2011 Jul 10;13(8):958-65. doi: 10.1038/ncb2286. PMID 21743466
- [Background] Zaragosi LE, Wdziekonski B, Brigand KL, Villageois P, Mari B, Waldmann R, Dani C, Barbry P. Small RNA sequencing reveals miR-642a-3p as a novel adipocyte-specific microRNA and miR-30 as a key regulator of human adipogenesis. Genome Biol. 2011 Jul 18;12(7):R64. doi: 10.1186/gb-2011-12-7-r64. PMID 21767385
- [Background] Meerson A, Traurig M, Ossowski V, Fleming JM, Mullins M, Baier LJ. Human adipose microRNA-221 is upregulated in obesity and affects fat metabolism downstream of leptin and TNF-alpha. Diabetologia. 2013 Sep;56(9):1971-9. doi: 10.1007/s00125-013-2950-9. Epub 2013 Jun 12. PMID 23756832
- [Background] Pasquinelli AE, Reinhart BJ, Slack F, Martindale MQ, Kuroda MI, Maller B, Hayward DC, Ball EE, Degnan B, Muller P, Spring J, Srinivasan A, Fishman M, Finnerty J, Corbo J, Levine M, Leahy P, Davidson E, Ruvkun G. Conservation of the sequence and temporal expression of let-7 heterochronic regulatory RNA. Nature. 2000 Nov 2;408(6808):86-9. doi: 10.1038/35040556. PMID 11081512
- [Background] Lagos-Quintana M, Rauhut R, Lendeckel W, Tuschl T. Identification of novel genes coding for small expressed RNAs. Science. 2001 Oct 26;294(5543):853-8. doi: 10.1126/science.1064921. PMID 11679670
- [Background] Lee RC, Ambros V. An extensive class of small RNAs in Caenorhabditis elegans. Science. 2001 Oct 26;294(5543):862-4. doi: 10.1126/science.1065329. PMID 11679672
- [Background] Lau NC, Lim LP, Weinstein EG, Bartel DP. An abundant class of tiny RNAs with probable regulatory roles in Caenorhabditis elegans. Science. 2001 Oct 26;294(5543):858-62. doi: 10.1126/science.1065062. PMID 11679671
- [Background] Filipowicz W, Bhattacharyya SN, Sonenberg N. Mechanisms of post-transcriptional regulation by microRNAs: are the answers in sight? Nat Rev Genet. 2008 Feb;9(2):102-14. doi: 10.1038/nrg2290. PMID 18197166
- [Background] Martinelli R, Nardelli C, Pilone V, Buonomo T, Liguori R, Castano I, Buono P, Masone S, Persico G, Forestieri P, Pastore L, Sacchetti L. miR-519d overexpression is associated with human obesity. Obesity (Silver Spring). 2010 Nov;18(11):2170-6. doi: 10.1038/oby.2009.474. Epub 2010 Jan 7. PMID 20057369
- [Background] Kloting N, Berthold S, Kovacs P, Schon MR, Fasshauer M, Ruschke K, Stumvoll M, Bluher M. MicroRNA expression in human omental and subcutaneous adipose tissue. PLoS One. 2009;4(3):e4699. doi: 10.1371/journal.pone.0004699. Epub 2009 Mar 4. PMID 19259271
- [Background] Herrera BM, Lockstone HE, Taylor JM, Ria M, Barrett A, Collins S, Kaisaki P, Argoud K, Fernandez C, Travers ME, Grew JP, Randall JC, Gloyn AL, Gauguier D, McCarthy MI, Lindgren CM. Global microRNA expression profiles in insulin target tissues in a spontaneous rat model of type 2 diabetes. Diabetologia. 2010 Jun;53(6):1099-109. doi: 10.1007/s00125-010-1667-2. Epub 2010 Mar 3. PMID 20198361
- [Background] Xie H, Lim B, Lodish HF. MicroRNAs induced during adipogenesis that accelerate fat cell development are downregulated in obesity. Diabetes. 2009 May;58(5):1050-7. doi: 10.2337/db08-1299. Epub 2009 Feb 2. PMID 19188425
- [Background] Turchinovich A, Samatov TR, Tonevitsky AG, Burwinkel B. Circulating miRNAs: cell-cell communication function? Front Genet. 2013 Jun 28;4:119. doi: 10.3389/fgene.2013.00119. Print 2013. PMID 23825476
- [Background] Ogawa R, Tanaka C, Sato M, Nagasaki H, Sugimura K, Okumura K, Nakagawa Y, Aoki N. Adipocyte-derived microvesicles contain RNA that is transported into macrophages and might be secreted into blood circulation. Biochem Biophys Res Commun. 2010 Aug 6;398(4):723-9. doi: 10.1016/j.bbrc.2010.07.008. Epub 2010 Jul 17. PMID 20621060
- [Background] Deng ZB, Poliakov A, Hardy RW, Clements R, Liu C, Liu Y, Wang J, Xiang X, Zhang S, Zhuang X, Shah SV, Sun D, Michalek S, Grizzle WE, Garvey T, Mobley J, Zhang HG. Adipose tissue exosome-like vesicles mediate activation of macrophage-induced insulin resistance. Diabetes. 2009 Nov;58(11):2498-505. doi: 10.2337/db09-0216. Epub 2009 Aug 12. PMID 19675137
- [Background] Dietze D, Koenen M, Rohrig K, Horikoshi H, Hauner H, Eckel J. Impairment of insulin signaling in human skeletal muscle cells by co-culture with human adipocytes. Diabetes. 2002 Aug;51(8):2369-76. doi: 10.2337/diabetes.51.8.2369. PMID 12145147
- [Background] Dietze-Schroeder D, Sell H, Uhlig M, Koenen M, Eckel J. Autocrine action of adiponectin on human fat cells prevents the release of insulin resistance-inducing factors. Diabetes. 2005 Jul;54(7):2003-11. doi: 10.2337/diabetes.54.7.2003. PMID 15983200
- See also: Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org